CLINICAL TRIAL: NCT00021697
Title: A Double-Blind Controlled, Multicenter Phase II/III Study to Assess the Safety and Efficacy of AVP-923 (Dextromethorphan/Quinidine) in the Treatment of Pseudobulbar Affect in Patients With Amyotrophic Lateral Sclerosis
Brief Title: Safety/Efficacy of AVP-923 in the Treatment of Emotional Lability (Uncontrolled Crying & Laughing) in Patients With ALS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Avanir Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 99-AVR-102; AVP-923
Record Dates: First submitted 2001-08-01; First posted 2001-08-03 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: AVP-923; Dextromethorphan; Quinidine; Pseudobulbar Affect
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — dextromethorphan - quinidine combination

INTERVENTIONS:
Drug: AVP-923

SUMMARY:
The purpose of this study is to compare and evaluate the safety of AVP-923 (dextromethorphan/quinidine) for the treatment of emotional lability in ALS patients.

ELIGIBILITY:
Inclusion:

* 18 to 80 years of age, inclusive
* Confirmed diagnosis of ALS or probable ALS
* Clinical history of pseudobulbar affect
* If female, must not be pregnant, breast-feeding, or planning a pregnancy during the course of the study, and must have a negative urine pregnancy test prior to start of study
* If female, must have been practicing an established method of birth control for at least the prior month (oral contraceptive tablets, hormonal implant device, intrauterine device, diaphragm and contraceptive cream or foam, condom with spermicide, tubal ligation, or abstinence) or be surgically sterile or post-menopausal
* Must be willing to not take any prohibited medications during participation in the study

Exclusion:

* Known sensitivity to quinidine or opiate drugs (codeine, etc.)
* On any anti-depressive medication
* Recently (within two months) diagnosed with ALS
* Currently participating in, or who within the past 30 days have participated in, the study of another investigational new drug
* Previously received treatment with co-administration of dextromethorphan and quinidine
* History of substance abuse within the past two years
* Women who are pregnant or likely to become pregnant during the course of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2001-01; Primary Completion 2002-04 (Actual); Study Completion 2002-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Loma Linda University Dept. of Neurology, Loma Linda, California
  - UCLA School of Medicine Dept. of Neurology, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado Health Sciences, Denver, Colorado
  - University of Miami Dept. of Neurology, Miami, Florida
  - Northwestern Medical School, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Columbia-Presbyterian Center Neurological Institute, New York, New York
  - State University of New York, Syracuse, New York
  - Carolinas Medical Center Carolinas Neuromuscular/ALS-MDA Center, Charlotte, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - MCP-Hahnemann University Dept. of Neurology, Philadelphia, Pennsylvania
  - Penn Neurological Institute, Philadelphia, Pennsylvania
  - University of Texas Health Science Center @ San Antonio, San Antonio, Texas
  - University of Wisconsin ALS Clinical Research Center, Madison, Wisconsin

REFERENCES:
- [Background] Dark FL, McGrath JJ, Ron MA. Pathological laughing and crying. Aust N Z J Psychiatry. 1996 Aug;30(4):472-9. doi: 10.3109/00048679609065020. PMID 8887697
- [Background] Smith RA, Moore SR, Gresham LS, Manley PE, Licht JM: The treatment of affective lability with dextromethorphan. Neurology 54: 604P, 1995
- [Background] Gallagher JP. Pathologic laughter and crying in ALS: a search for their origin. Acta Neurol Scand. 1989 Aug;80(2):114-7. doi: 10.1111/j.1600-0404.1989.tb03851.x. PMID 2816272
- [Background] Wolf JK, Santana HB, Thorpy M. Treatment of "emotional incontinence" with levodopa. Neurology. 1979 Oct;29(10):1435-6. doi: 10.1212/wnl.29.10.1435-b. No abstract available. PMID 573397
- [Background] Muller U, Murai T, Bauer-Wittmund T, von Cramon DY. Paroxetine versus citalopram treatment of pathological crying after brain injury. Brain Inj. 1999 Oct;13(10):805-11. doi: 10.1080/026990599121197. PMID 10576464
- [Background] Moore SR, Gresham LS, Bromberg MB, Kasarkis EJ, Smith RA. A self report measure of affective lability. J Neurol Neurosurg Psychiatry. 1997 Jul;63(1):89-93. doi: 10.1136/jnnp.63.1.89. PMID 9221973
- [Background] Schadel M, Wu D, Otton SV, Kalow W, Sellers EM. Pharmacokinetics of dextromethorphan and metabolites in humans: influence of the CYP2D6 phenotype and quinidine inhibition. J Clin Psychopharmacol. 1995 Aug;15(4):263-9. doi: 10.1097/00004714-199508000-00005. PMID 7593709
- [Background] Brooks BR, Crumpacker D, Fellus J, Kantor D, Kaye RE. PRISM: a novel research tool to assess the prevalence of pseudobulbar affect symptoms across neurological conditions. PLoS One. 2013 Aug 21;8(8):e72232. doi: 10.1371/journal.pone.0072232. eCollection 2013. PMID 23991068
- [Result] Brooks BR, Thisted RA, Appel SH, Bradley WG, Olney RK, Berg JE, Pope LE, Smith RA; AVP-923 ALS Study Group. Treatment of pseudobulbar affect in ALS with dextromethorphan/quinidine: a randomized trial. Neurology. 2004 Oct 26;63(8):1364-70. doi: 10.1212/01.wnl.0000142042.50528.2f. PMID 15505150
- See also: Homepage for ALSA/ALS — http://www.alsa.org